CLINICAL TRIAL: NCT06743256
Title: Prospective, Multi-center, Single-arm, Open Label Study Designed to Assess the Safety and Feasibility of the Levita Magnetic Surgical System in Laparoscopic Gynecological Procedures
Brief Title: Study Designed to Assess the Safety and Feasibility of the Levita Magnetic Surgical System in Laparoscopic Gynecological Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Levita Magnetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LVT010
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Gynecological Laparoscopic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Magnetic Surgical System in laparoscopic gynecological procedures (Experimental)
  Interventions: Device: Surgical System

INTERVENTIONS:
Device: Surgical System — Levita Magnetic Surgical System

SUMMARY:
A study at multiple centers to evaluate the safety and practicality of the Levita Magnetic Surgical System for use in laparoscopic gynecological surgeries.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Having a BMI of at least 20 kg/m2
* Scheduled to undergo elective gynecological procedure
* Willing and able to provide a written Informed Consent Form (ICF) to participate in the study prior to any study required procedures

Exclusion Criteria:

* Individuals with BMI higher than 60 kg/m2.
* Emergency procedures (e.g., ectopic pregnancy, severe bleeding).
* Significant comorbidities: e.g. cardiovascular, neuromuscular, chronic obstructive pulmonary disease, and urological disease (renal failure).
* Individuals with pacemakers, defibrillators, or other electromedical implants.
* Individuals with ferromagnetic implants.
* Clinical history of impaired coagulation confirmed by abnormal blood tests.
* Anatomical abnormality or disease of intended target tissue noted after initiation of index procedure that would prevent device use.
* Pregnant or wishes to become pregnant during the length of study participation.
* Individual is not likely to comply with the follow-up evaluation schedule.
* Participating in a clinical trial of another investigational drug or device.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Enrollment: 50 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-05-07 (Estimated); Study Completion 2026-06-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Device and/or Procedure Related Adverse Events | From enrollment to end of follow up at 30 days.
  Adverse events will be summarized by relatedness to the device and/or procedure, seriousness and level of severity.
Average Number of Ports | During index procedure.
  Ability to adequately retract the uterus, adnexal organs, and peri uterine tissue to achieve an effective exposure of the target tissue.
  Adequate retraction will be deemed to be achieved if an additional port that is typically used for retraction and exposure of target tissues can be eliminated.

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - Hospital Clinico San Borja Arriaran, Peñalolén, Santiago Metropolitan
  - Hospital Santiago Oriente "Dr. Luis Tisné Brousse", Peñalolén, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: Undecided